CLINICAL TRIAL: NCT05733000
Title: Phase II Open-Label Multi-Cohort Study Evaluating CPI-613 (Devimistat) in Combination With Hydroxychloroquine and 5-fluorouracil or Gemcitabine in Patients With Advanced Chemorefractory Colorectal, Pancreatic, or Other Solid Cancers
Brief Title: CPI-613 (Devimistat) in Combination With Hydroxychloroquine and 5-fluorouracil or Gemcitabine in Treating Patients With Advanced Chemorefractory Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 22MH03; NCI-2023-00070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00218203 (Other: Northwestern IRB); NU 22MH03 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-17 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Advanced Biliary Tract Carcinoma; Advanced Colorectal Carcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Advanced Lung Adenocarcinoma; Advanced Malignant Solid Neoplasm; Advanced Ovarian Carcinoma; Advanced Pancreatic Carcinoma; Advanced Urothelial Carcinoma; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Biliary Tract Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Lung Adenocarcinoma; Metastatic Ovarian Carcinoma; Metastatic Pancreatic Carcinoma; Metastatic Urothelial Carcinoma; Refractory Biliary Tract Carcinoma; Refractory Colorectal Carcinoma; Refractory Gastroesophageal Junction Adenocarcinoma; Refractory Lung Adenocarcinoma; Refractory Ovarian Carcinoma; Refractory Pancreatic Carcinoma; Refractory Urothelial Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma of Lung; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Transitional Cell; Lung Neoplasms | interventions — Specimen Handling; devimistat; Fluorouracil; dehydroftorafur; Gemcitabine; Hydroxychloroquine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- COHORT 1 (Devimistat, 5-FU, HCQ) (Experimental): Patients with colorectal cancer receive devimistat IV, 5-FU IV, plus HCQ PO on study. Patients also undergo CT and/or MRI and undergo blood specimen collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Devimistat; Drug: Fluorouracil; Drug: Hydroxychloroquine; Procedure: Magnetic Resonance Imaging
- COHORT 2 (Devimistat, 5-FU, HCQ) (Experimental): Patients with pancreatic cancer receive devimistat IV, 5-FU IV, plus HCQ PO on study. Patients also undergo CT and/or MRI and undergo blood specimen collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Devimistat; Drug: Fluorouracil; Drug: Hydroxychloroquine; Procedure: Magnetic Resonance Imaging
- COHORT 3 (Devimistat, 5-FU, HCQ, Gemcitabine) (Experimental): Patients with gastroesophageal cancer receive devimistat IV, 5-FU IV, plus HCQ PO on study. Patients with urothelial, ovarian, or non-small cell lung cancer receive devimistat IV, gemcitabine IV, plus HCQ PO on study. Patients with biliary tumors receive devimistat IV and gemcitabine IV or HCQ PO on study. Patients also undergo CT and/or MRI and undergo blood specimen collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Devimistat; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Drug: Hydroxychloroquine; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Devimistat — Receive IV
  Other Names: Alpha-Lipoic Acid Analogue CPI-613; CPI 613; CPI-613
Drug: Fluorouracil — Receive IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine Hydrochloride — Receive IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
  Arms: COHORT 3 (Devimistat, 5-FU, HCQ, Gemcitabine)
Drug: Hydroxychloroquine — Receive PO
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase II trial tests how well CPI-613 (devimistat) in combination with hydroxychloroquine (HCQ) and 5-fluorouracil (5-FU) or gemcitabine works in patients with solid tumors that may have spread from where they first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that have not responded to chemotherapy medications (chemorefractory). Metabolism is how the cells in the body use molecules (carbohydrates, fats, and proteins) from food to get the energy they need to grow, reproduce and stay healthy. Tumor cells, however, do this process differently as they use more molecules (glucose, a type of carbohydrate) to make the energy they need to grow and spread. CPI-613 works by blocking the creation of the energy that tumor cells need to survive, grow in the body and make more tumor cells. When the energy production they need is blocked, the tumor cells can no longer survive. Hydroxychloroquine is a drug used to treat malaria and rheumatoid arthritis and may also improve the immune system in a way that tumors may be better controlled. Fluorouracil is in a class of medications called antimetabolites. It works by killing fast-growing abnormal cells. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill tumor cells. CPI-613 (devimistat) in combination with hydroxychloroquine and 5-fluorouracil or gemcitabine may work to better treat advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The primary objective of this study will be to estimate the overall response rate (ORR) of treatment with devimistat (CPI-613) plus HCQ and, depending on the cohort and indication, either 5-FU or gemcitabine.

SECONDARY OBJECTIVES:

I. Evaluate progression-free survival (PFS) of patients with solid tumors that are treated with CPI-613 plus HCQ and, depending on the cohort and indication, either 5-FU or gemcitabine.

II. Determine overall survival (OS) of patients with solid tumors that are treated with CPI-613 plus HCQ and, depending on the cohort and indication, either 5-FU or gemcitabine.

III. Assess duration of response (DOR) of patients with solid tumors that are treated with CPI-613 plus HCQ and, depending on the cohort and indication, either 5-FU or gemcitabine.

IV. Assess safety and tolerability for patients with solid tumors treated with specified treatments.

EXPLORATORY OBJECTIVES:

I. Blood from patients in cohort 3 that consent will be collected at baseline, cycle 1, day 1 (C1D1), C1D15, C2D1, and at the time of treatment discontinuation for further molecular and metabolic analysis, possibly including but not limited to proteomic, metabolomic, and genetic/genomic analysis.

OUTLINE: Patients are assigned to 1 of 3 cohorts.

COHORT 1: Patients with colorectal cancer receive devimistat intravenously (IV), 5-FU IV, plus HCQ orally (PO) on study. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) and undergo blood specimen collection throughout the study.

COHORT 2: Patients with pancreatic cancer receive devimistat IV, 5-FU IV, plus HCQ PO on study. Patients also undergo CT and/or MRI and undergo blood specimen collection throughout the study.

COHORT 3: Patients with gastroesophageal cancer receive devimistat IV, 5-FU IV, plus HCQ PO on study. Patients with urothelial, ovarian, or non-small cell lung cancer receive devimistat IV, gemcitabine IV, plus HCQ PO on study. Patients with biliary tumors receive devimistat IV and gemcitabine IV or HCQ PO on study. Patients also undergo CT and/or MRI and undergo blood specimen collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed cancer for which standard-of-care curative measures are no longer effective or be intolerant to those agents. Patients in cohort 1 must have colorectal cancer. Patients in cohort 2 must have pancreatic cancer. Patients in cohort 3 may have any of the following cancers:

  * Biliary
  * Gastroesophageal
  * Urothelial
  * Ovarian
  * Non-small cell lung (adenocarcinoma only)
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 disease.
* Patients must have radiographic documentation of metastatic disease with imaging within =< 6 weeks prior to registration.
* Patients must be age >= 18 years.
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. Performance Status of 2 will be allowed with approval from principle investigator (PI) on a case-by case basis.

  * Note: Performance status of 2 will be allowed with approval from PI on a case-by case basis. Documentation of PI approval in these cases will be stored with inclusion/exclusion signed checklist for patient and/or in patient's shadow chart.
* Patients must have exhausted all available molecularly targeted therapies (e.g., anti-PD-1/anti-PD-L1 agents where indicated).
* Absolute neutrophil count (ANC) >= 1,500/mcL (within the last 14 days of screening)
* Hemoglobin (Hgb) >= 9 g/dL (within the last 14 days of screening) (Transfusions permitted. Eligibility labs should be drawn >= 7 days from transfusion).
* Platelets (PLT) >= 100,000/mcL (within the last 14 days of screening) (Transfusions permitted. Eligibility labs should be drawn >= 7 days from transfusion).
* INR (international normalized ratio) =< 1.6 (within the last 14 days of screening) (unless receiving anticoagulation therapy) If receiving anticoagulant: INR =< 3.0 and no active bleeding, (i.e., no bleeding within 14 days prior to first dose of study therapy).
* Total bilirubin =<1.5 x Institutional upper limit of normal (ULN) (within the last 14 days of screening)

  * Note: Patients with Gilbert's Syndrome are exempt. Patients with liver metastases with no significant bilirubin obstruction may have a total bilirubin level of =< 2.0 mg/dL.
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) =< 2.5 x institutional ULN (within the last 14 days of screening)

  * Note: If liver metastases are present, then =< 5 x ULN is allowed.
* Alanine transaminase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 2.5 x institutional ULN (within the last 14 days of screening)

  * Note: If liver metastases are present, then =< 5 x ULN is allowed.
* Serum albumin > 3.0 g/dL (within the last 14 days of screening)
* Creatinine =< 1.5 x ULN OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (within the last 14 days of screening)

  * eGFR is estimated GFR calculated by the abbreviated Modification of Diet in Renal Disease (MDRD) equation
* The effects of combination treatment of CPI-613, 5-FU, gemcitabine, and HCQ on the developing human fetus are unknown. For this reason and because antineoplastic agents as well as other therapeutic agents used in this trial are known to be teratogenic, patients of child-bearing potential (POCBP) regardless of gender must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 180 days following completion of therapy. Patients who can impregnate their partners regardless of gender must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 180 days following completion of therapy. Should a patient become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform their treating physician immediately.

  * Note: At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Note: A POCBP is any person with an egg-producing reproductive tract (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative pregnancy test prior to registration on study.

  * Note: If negative pregnancy test result is >7 days from first dose of study treatment it must be repeated at time of first dose of study treatment (with any of the four drugs used in this study).
* For patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration.
* For patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment, must have an undetectable HCV viral load. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardio toxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. Patients must be class 2B or better.

  * Note: Patients with pacemakers where corrected QT interval (QTc) is not a reliable measure will require an evaluation by a cardiologist to exclude co-existing cardiac conditions which would prohibit safe participation in the study.
* Patients must have the ability to understand and the willingness to sign a written informed consent document for the duration of the entirety of the study.
* Patients must be reliable, willing to make themselves available for the duration of the entire study and willing to follow screening procedures.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1).

  * Note: Patients who experience adverse events of alopecia and peripheral neuropathy that have not recovered are eligible; patients with any lab abnormality that is above grade 1 related to previous therapy found to be not clinically significant will also be eligible.
* Patients with symptomatic brain metastases currently using corticosteroids.

  * Note: Patients with brain metastases who are asymptomatic and off corticosteroids for at least one week are eligible.
* Patients with severe obstructive pulmonary disease or interstitial lung disease.
* Patients with a history of myocardial infarction that is <90 days prior to registration.
* Patients using concomitant medications that prolong the QT/QTc intervals. For example, patients receiving amiodarone. Using amiodarone together with hydroxychloroquine can increase the risk of long QT syndrome that although rare, may be serious, and potentially life-threatening.
* Patients with a history of additional risk factors for drug-induced QT prolongation or Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome).
* Patients with major surgery or significant traumatic injury =< 21 days prior to registration.
* Patients receiving treatment with low dose chemotherapy concurrent with radiation =< 21 days prior to registration.

OR patients who have had chemotherapy or radiotherapy =< 21 days (42 days for nitrosoureas or mitomycin C) prior to registration.

* Note: Palliative radiation before and during study participation is permissible providing it is not to a target lesion.

  * Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:
* Ongoing or active infection requiring systemic treatment.
* Clinically significant complications such as perforation, gastrointestinal bleeding, or diverticulitis within 42 days prior to registration.
* Symptomatic congestive heart failure; symptomatic coronary artery disease, symptomatic angina pectoris, or symptomatic myocardial infarction.
* Unstable angina pectoris.
* Unstable cardiac arrhythmia.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Active substance abuse.
* Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.

  * Patients who are pregnant or nursing.
  * Patients with Fridericia-corrected QT interval (QTcF) > 470 msec (female) or > 450 (male), or history of congenital long QT syndrome. Any electrocardiogram (ECG) abnormality that in the opinion of the investigator would preclude safe participation in the study.
  * Patients who have pre-existing retinopathy of the eye.
  * Patients who are unable to swallow or retain and absorb oral medication
  * Patients with known hypersensitivity to any of the following: CPI or its inactive components, 4-aminoquinoline compounds, or quinine.
  * Patients with poorly controlled diabetes mellitus (glycosylated hemoglobin (HbA1c) of > 7%, pre-prandial capillary plasma glucose > 130mg/dl, and peak postprandial capillary plasma glucose of > 180mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2028-01-04 (Estimated); Study Completion 2030-03-04 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Time from baseline to disease progression, initiates subsequent anti-cancer therapy, or 24 months (whichever occurs first)
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 in patients with solid tumors treated under this protocol. ORR is defined as the percentage of patients with documented complete response (CR) plus the percentage of patients with documented partial response (PR). ORR will be reported with the corresponding exact confidence intervals.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time that elapses between the day of subject registration and the earlier of the day of first documented disease progression by clinical or radiographic evaluation or death from any cause, assessed up to 24 months
  Will be assessed using Kaplan-Meier estimates. PFS for the main cohorts (cohort 1 and cohort 2) and exploratory cohort (cohort 3) will be analyzed and reported separately.
Overall survival (OS) | Time that elapses between the day of subject registration and death from any cause, assessed up to 24 months
  Will be assessed using Kaplan-Meier estimates. OS for the main cohort and exploratory cohort will be analyzed and reported separately.
Duration of response (DOR) | Time elapsed from the day when CR or PR is first observed until the earlier of the day of first documented disease progression or death, assessed up to 24 months
  Will be assessed using Kaplan-Meier estimates. DOR for the main cohorts and exploratory cohort will be analyzed and reported separately.
Incidence of adverse events | Up to 30 days post treatment
  Will be assessed using the National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States